CLINICAL TRIAL: NCT01171716
Title: The Body's Response to Changes in Dietary Protein and Meal-Frequency In Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Purdue University (Other)
Responsible Party: Principal Investigator, Wayne Campbell, Wayne Campbell, Ph. D, Purdue University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 0708005744
Record Dates: First submitted 2010-07-27; First posted 2010-07-28 (Estimated); Last update posted 2013-01-17 (Estimated); Status verified 2013-01

CONDITIONS: Low Protein Dietary Intake; High Protein Dietary Intake
Keywords: overweight, protein intake, satiety, eating, meal patterns
MeSH Terms: conditions — Overweight

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dietary Protein Intake (Other): LP intake 3 meals and 6 meals HP intake 3 meals and 6 meals
  Interventions: Other: Meal Patterning

INTERVENTIONS:
Other: Meal Patterning — LP intake 3 meals and 6 meals HP intake 3 meals and 6 meals

SUMMARY:
the purpose of this study is to identify how the body responds to increased dietary protein (that includes pork and eggs) and meal-frequency in adult men. During this study, the changes in blood glucose, hormones, appetite, and energy expenditure will be examined.

ELIGIBILITY:
Inclusion Criteria:

* 21 and older, BMI between 25.0-34.6, Weight Stable for at least 6 mths, body >25%, non smoking, clinically normal blood profiles, non-diabetic.

Exclusion Criteria:

* intermittently been involved in a diet and/or exercise program within the last 3 months, Have no allergies to eggs.

Min Age: 21 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2007-09; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
The Body's Response to Changes in Dietary Protein and Meal-Frequency In Men | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Purdue University, Dept of Foods and Nutrition, West Lafayette, Indiana, United States